CLINICAL TRIAL: NCT00761163
Title: The Body's Response to Aerobic Versus Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Wayne Campbell, Ph. D., Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0701004892; NIH/NIA 5R01AG021911
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Exercise
Keywords: The purpose of this study is to identify the body's response to aerobic vs. resistance exercise
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training; Exercise

ARMS (3):
- 1 (Experimental)
  Interventions: Other: Resistance Exercise
- 2 (Experimental)
  Interventions: Other: Aerobic Exercise
- 3 (Experimental)
  Interventions: Other: Control (Non-exercise)

INTERVENTIONS:
Other: Resistance Exercise — The subjects will complete 2 resistive exercise sessions on non-consecutive days that will be supervised by our laboratory staff. The following exercises will be performed using the Keiser Sports Health equipment in Ismail Health, Exercise, and Nutrition Center: seated row, double leg press, seated leg curl, chest press, and leg extension. The subjects will individually perform 3 sets of 8-10 repetitions at an exercise intensity of 70% of pre-determined maximal strength for these exercises. Each repetition will be performed in a slow (six to eight seconds) uniform fashion, giving equal time to the concentric (muscle shortening) and eccentric (muscle lengthening) portions. One minute of rest will be allowed between sets. The last repetition of the third set of each exercise will be done to voluntary fatigue or the performance of 12 repetitions.
  Arms: 1
Other: Aerobic Exercise — The subjects will complete 2 aerobic exercise sessions on non-consecutive days that will also be supervised by our laboratory staff. The subjects will perform 45 minutes of aerobic exercise on a stationary bike at an exercise intensity of 70% of their heart-rate reserve.
  Arms: 2
Other: Control (Non-exercise) — The subjects will also complete 2 non-exercise sessions on non-consecutive days that will also be supervised by our laboratory staff. These sessions will consist of incorporating diversionary tasks throughout a 45 minute period consisting of a variety of motor and psychological tasks (tests of hand steadiness, alertness, optical illusions, mental acuity, etc.)
  Arms: 3

SUMMARY:
The purpose of this study is to identify the body's response to aerobic vs. resistance exercise. Throughout this study, we will examine food intake, appetite, and physical and mental well-being before, during, and after aerobic and resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18-29 kg/m2
* Weight stable (< 4.5 kg weight change within last 6 months)
* Non-smoking
* Constant habitual activity patterns within last 3 months
* Non-diabetic
* Resistive exercise training (≥ 2 times a week) based on reported physical activity levels (questionnaire)
* Aerobic exercise training (≥ 2 times a week, 30-min sessions) based on reported physical activity levels (questionnaire)
* Confirmation of acceptability of eating the study test foods (macaroni casserole)
* Approved to participate in this study by our study physician and principle investigator

The older subjects must also meet the following eligibility criteria:

* Age range: 65 years and older
* Body fat (women: <38%; men: <28%)
* Normal resting EKG as assessed by a Cardiologist

The younger subjects must also meet the following eligibility criteria:

* Age range: 18-29 years
* Body fat (women: <28%; men: <18%)

Exclusion Criteria:

* Body mass index: outside of the 18-29 kg/m2 range
* Gained or lost > 4.5 kg within the last 6 months
* Smoker (currently or within the last year)
* Intermittently been involved in a diet and/or exercise program within the last 3 months
* Clinically diagnosed as diabetic
* Did not perform resistive exercise training (currently or within the last 3 months) based on reported physical activity levels (questionnaire)
* Did not perform adequate aerobic exercise (currently or within the last 3 months) based on physical activity levels (questionnaire)
* Study food is found to be unacceptable for consumption by the subject
* Unapproved to participate in this study by our study physician and principle investigator

The older subjects:

* Age range: <65 yrs
* Body fat (women: >38%; men: >28%)
* Abnormal resting EKG (interpreted by a cardiologist) and assessed (for study exclusion) by our study physician, Arthur Rosen, MD

The younger subjects:

* Age range: outside the >29 yrs or <18 yrs
* Body fat (women: >28%; men: >18%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Physical well being via electrocardiogram and body composition | 5-6 weeks
Mental well being via questionnaires | 5-6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Laan DJ, Leidy HJ, Lim E, Campbell WW. Effects and reproducibility of aerobic and resistance exercise on appetite and energy intake in young, physically active adults. Appl Physiol Nutr Metab. 2010 Dec;35(6):842-7. doi: 10.1139/H10-072. PMID 21164556